CLINICAL TRIAL: NCT06567743
Title: A Phase 2, Multi-Arm, Multi-Cohort, Open-Label Study to Evaluate the Safety and Efficacy of Cretostimogene Grenadenorepvec in Participants With High-Risk Non-Muscle-Invasive Bladder Cancer (NMIBC)
Brief Title: Phase 2 Study to Evaluate Safety and Efficacy of Cretostimogene Grenadenorepvec in High-Risk NMIBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CG Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORE-008
Record Dates: First submitted 2024-08-14; First posted 2024-08-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: High-Risk Non-Muscle-Invasive Bladder Cancer
Keywords: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Experimental: Cohort A, Arm 1 (Experimental): Cretostimogene (1 x 1012 vp) will be administered intravesically via the current instillation method
  Interventions: Drug: Cretostimogene Grenadenorepvec
- Experimental: Cohort A, Arm 2 (Experimental): Cretostimogene (1 x 1012 vp) will be administered intravesically via an alternative instillation method.
  Interventions: Drug: Cretostimogene Grenadenorepvec
- Experimental: Cohort A, Arm 3 (Experimental): Cretostimogene (1 x 1012 vp) will be administered intravesically via an alternative instillation method.
  Interventions: Drug: Cretostimogene Grenadenorepvec
- Experimental: Cohort B, Arm 1 (Experimental): Cretostimogene (1 x 1012 vp) will be administered intravesically via an alternative instillation method.
  Interventions: Drug: Cretostimogene Grenadenorepvec
- Experimental: Cohort B, Arm 2 (Experimental): Cretostimogene (1 x 1012 vp) will be administered intravesically via an alternative instillation method.
  Interventions: Drug: Cretostimogene Grenadenorepvec
- Experimental: Cohort CX, Arm 1 (Experimental): At all treatment visits cretostimogene (1 x 1012 vp) will be administered intravesically via an alternative instillation method followed by gemcitabine instilled intravesically
  Interventions: Drug: Cretostimogene Grenadenorepvec
- Experimental: Cohort CX, Arm 2 (Experimental): Cretostimogene (1 x 1012 vp) will be administered intravesically via an alternative instillation method for two consecutive weeks, followed by gemcitabine administered intravesically in the third week on a cyclic 2:1 visit schedule basis
  Interventions: Drug: Cretostimogene Grenadenorepvec

INTERVENTIONS:
Drug: Cretostimogene Grenadenorepvec — Respective Cohort
  Other Names: CG0070

SUMMARY:
This is a Phase 2, Multi-Arm, Multi-Cohort, Open-Label Study to Evaluate the Safety and Efficacy of Cretostimogene Grenadenorepvec in Participants with High-Risk Non-Muscle-Invasive Bladder Cancer.

DETAILED DESCRIPTION:
In Cohort A, up to 125 participants will be enrolled with pathologically confirmed, high-risk high-grade non-muscle invasive bladder cancer (NMIBC) NMIBC (i.e., CIS with or without concomitant Ta or T1 disease OR HG Ta/T1 disease without CIS) which is naïve to Bacillus Calmette-Guerin (BCG) treatment. Participants with CIS with or without concomitant Ta/T1 NMIBC at baseline will be randomized 1:1 to receive cretostimogene via the current (Arm 1) or an alternative instillation procedure (Arm 2). Participants with papillary-only high-risk NMIBC (i.e., HG Ta/T1 without CIS) at baseline (Arm 3) will receive cretostimogene via the alternative instillation procedure.

In Cohort B, up to 150 participants will be enrolled with pathologically confirmed, high-risk high-grade NMIBC (i.e., CIS with or without concomitant Ta or T1 disease OR HG Ta/T1 disease without CIS) which has previously been exposed to BCG treatment. Participants with CIS-containing pathology at baseline will be recruited into Arm 1 and participants with papillary-only pathology at baseline will be recruited into Arm 2. Both Cohort B Arms 1 and 2 will receive cretostimogene via the alternative instillation procedure.

In Cohort CX, up to 50 participants will be enrolled with pathologically confirmed, high-risk high-grade NMIBC (i.e., CIS with or without concomitant Ta or T1 disease OR HG Ta/T1 disease without CIS) which has previously been exposed to or is unresponsive to BCG treatment. Participants will be randomized 1:1 to receive cretostimogene and gemcitabine either concurrently or sequentially.

In all cohorts, study treatment will be administered as a weekly induction course for the first 6 weeks with a reinduction course administered to patients who have CIS and/or high-grade Ta disease at the 3-month evaluation. Following induction, if no high-grade disease is detected, maintenance treatment will begin. This consists of a cycle of three weekly treatments every three months during the first year, and every six months during the second year, with an optional extension to the third year following the same six-month schedule.

Disease status will be assessed using urine cytology, complete bladder visualization (e.g., cystoscopy), upper tract assessment and directed resection/biopsy (if indicated) every 3 months for the first 2 years and then every 6 months for a further 2 years or until disease recurrence.

ELIGIBILITY:
Cohort A Key Inclusion Criteria:

* Pathologically confirmed BCG-naïve high-risk high-grade NMIBC (i.e., CIS with or without Ta/T1 disease or high-grade Ta/T1 papillary-only disease without CIS) within 90 days of treatment allocation.
* All visible disease must be resected, and all CIS resected or fulgurated, as feasible within 90 days prior to treatment allocation.
* Acceptable baseline organ function.

Cohort B Key Inclusion Criteria:

* Pathologically confirmed BCG-exposed high-risk high-grade NMIBC (i.e., CIS with or without Ta/T1 disease or high-grade Ta/T1 papillary-only disease without CIS) within 90 days of treatment allocation.
* All visible disease must be resected, and all CIS resected or fulgurated, as feasible within 90 days prior to treatment allocation.
* Acceptable baseline organ function.

Cohort CX Inclusion Criteria

* Pathologically confirmed high-risk high-grade BCG-unresponsive or BCG-exposed NMIBC (i.e., CIS with or without Ta/T1 disease or high-grade Ta/T1 papillary-only disease without CIS) within 90 days of treatment allocation.
* All visible disease must be resected, and all CIS resected or fulgurated, as feasible within 90 days prior to treatment allocation.
* Acceptable baseline organ function.

Key Exclusion Criteria (Both Cohorts):

* Current or past history of muscle-invasive, locally advanced or metastatic bladder cancer.
* High-grade urothelial carcinoma in the upper urinary tract or prostatic urethra within 24 months or T2 in upper tract within 48 months or any history of locally advanced/ nodal or metastatic disease in the upper urinary tract.
* Significant immunodeficiency.
* Pregnant or breastfeeding.
* Cohort CX Only: serial intravesical gemcitabine within 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Cohort A (Arm 1 and 2): Complete response rate | At 11 and 24 weeks
  Determine the complete response rate at any time following treatment with cretostimogene in participants with BCG-naïve CIS with or without concomitant high-grade Ta or T1 disease at baseline
Cohort A (Arm 3): High- Grade Event-Free Survival | 48 months
  Determine the High-Grade Event-Free Survival following treatment with cretostimogene in participants with BCG-naïve HG Ta/T1 disease without concomitant CIS at baseline.
Cohort B (Arm 1): Complete response rate | At 11 and 24 weeks
  Determine the complete response rate at any time following treatment with cretostimogene in participants with BCG-exposed CIS with or without concomitant high-grade Ta or T1 disease at baseline.
Cohort B (Arm 2): High-Grade Event-Free Survival | 48 months
  Determine the High-Grade Event-Free Survival following treatment with cretostimogene in participants with BCG-exposed high-grade Ta/T1 papillary disease without CIS at baseline.
Cohort CX (Arms 1 and 2): High-Grade Event-Free Survival | 48 months
  Determine the High-Grade Event-Free Survival following treatment with cretostimogene in participants with BCG-exposed or BCG-unresponsive high-grade NMIBC.
Cohort CX (Arms 1 and 2): Safety | 48 months
  Determine the safety of concurrent cretostimogene and gemcitabine and sequential cretostimogene and gemcitabine.

SECONDARY OUTCOMES:
Cohort A (Arms 1 and 2): Evaluate cretostimogene instillation methods | At 11 and 24 weeks
  Evaluate cretostimogene genome and GM-CSF levels, treatment efficacy, and safety by 2 different methods of cretostimogene instillation in participants with pathologically confirmed CIS-containing high-risk NMIBC who are naïve to BCG treatment.
Cohort A (Arm 3): High-Grade Event-Free Survival at 12 months | At 12 months
  Determine the proportion of participants with BCG-naive papillary-only high-grade NMIBC at baseline who are free from high-grade events at 12 months
Cohort A (Arms 1 and 2) and Cohort B (Arm 1) Duration of response | 48 months
  Assess duration of response in participants with CIS with or without concomitant HG Ta/T1 disease at baseline
Cohort B (Arm 2) High-Grade Event-Free Survival at 12 months | At 12 months
  Determine the proportion of participants with BCG-exposed papillary-only high-grade NMIBC at baseline who are free from high-grade events at 12 months
Cohort CX (Arm 1 and 2) Complete response rate | At 11 and 24 weeks
  Determine the complete response rate at any time following treatment with cretostimogene and gemcitabine in participants with BCG-exposed or BCG-unresponsive CIS with or without concomitant high-grade Ta or T1 disease at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Kasturi, MD, Study Director — CG Oncology
Locations (65):
- United States (65):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arizona Urology Specialty, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Arkansas Urology, Little Rock, Arkansas
  - Michael G Oefelein, MD Clinical Trials, Bakersfield, California
  - Genesis Research (Greater Los Angeles), Los Alamitos, California
  - Advanced Urology, Los Angeles, California
  - Urology Center of Southern California, Murrieta, California
  - University of California, Irvine, Orange, California
  - Om research, San Diego, California
  - University of Southern California, San Diego, California
  - Genesis Research (Greater Los Angeles), Torrance, California
  - Colorado Urology, Lakewood, Colorado
  - Urology Associates, Lone Tree, Lone Tree, Colorado
  - University of Florida, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Advanced Urology Institute (Solaris), Largo, Florida
  - Advanced Urology Institute, Oxford, Florida
  - Advanced Urology Institute - Tallahassee (Solaris), Tallahassee, Florida
  - Emory University, Atlanta, Georgia
  - Associated Urological Specialists, Chicago Ridge, Illinois
  - Uropartners, Glenview, Illinois
  - Urology of Indiana - Carmel, Carmel, Indiana
  - Urology of Indiana, LLC (US Urology Partners), Greenwood, Indiana
  - First Urology, PSC, Jeffersonville, Indiana
  - Urologic Specialists of Northwest Indiana (Solaris), Merrillville, Indiana
  - Urology Center of Iowa Research, Clive, Iowa
  - Wichita Urology Group, Wichita, Kansas
  - Southern Urology (Urology America), Lafayette, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Anne Arundel Urology, Annapolis, Maryland
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Comprehensive Urology, Royal Oak, Michigan
  - Michigan Institute of Urology (Solaris), Troy, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Minnesota Urology, Woodbury, Minnesota
  - Specialty Clinical Research of St. Louis, St Louis, Missouri
  - Adult and Adolescent Urology, Omaha, Nebraska
  - Integrated Medical Professionals, PLLC (Solaris), New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Upstate, Syracuse, New York
  - Associated Medical Professionals of NY, PLLC (US Urology Partners), Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Urology Group (Solaris), Cincinnati, Ohio
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Central Ohio Urology Group (US Urology Partners), Gahanna, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - Midlantic Urology (Solaris), Bala-Cynwyd, Pennsylvania
  - Penn State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Charleston Area Medical Center, Charleston, South Carolina
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Lowcountry Urology (Solaris), North Charleston, South Carolina
  - The Conrad Pearson Clinic (Urology America), Germantown, Tennessee
  - Urology Associates, PC, Nashville, Tennessee
  - Amarillo Urology Research, Amarillo, Texas
  - UPNT Research Institute, LLC, Arlington, Texas
  - Urology Austin, PLLC (Urology America), Austin, Texas
  - Urology Clinics of North Texas, PLLC, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - Urology San Antonio, PA dba USA Clinical Trials, San Antonio, Texas
  - Urology of Virginia, Virginia Beach, Virginia
  - Spokane Urology, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No